CLINICAL TRIAL: NCT02968251
Title: Designing and Evaluating a School-based Hand Washing Program in Malawi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSEARS20160619001
Record Dates: First submitted 2016-10-11; First posted 2016-11-18 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2016-10

CONDITIONS: School-based, Hand-washing, Program, Malawi

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hand Washing Program (HWP) (Experimental): Clusters in this arm will be given a Hand Washing Program (HWP) which will consist of: integrating hand washing practice in the school health policy, setting up proper hand washing facilities in the intervention schools, training to school teachers, delivering of health talk to schoolchildren and their parents, developing reminders and posters of a simplified 5-step hand washing technique, peer briefing session, take home package (5-steps hand washing, commitment letter, poster, leaflet). The program will be delivered once every week.
  Interventions: Behavioral: Hand Washing Program (HWP)
- No Hand Washing Program (NHWP) (No Intervention): Clusters in this arm will be allowed to continue with their usual practice regarding hand washing/hygiene

INTERVENTIONS:
Behavioral: Hand Washing Program (HWP) — HWP consists of integrating hand washing practice in the school health policy, setting up proper hand washing facilities in the intervention schools, training to school teachers, delivering of health talk to schoolchildren and their parents, developing reminders and posters of a simplified 5-step hand washing technique, peer briefing session, take home package (5-steps hand washing, commitment letter, poster, leaflet). The program will be delivered once every week.
  Arms: Hand Washing Program (HWP)

SUMMARY:
The aim of the study is to design and evaluate a school-based hand washing program for children in Malawi, Sub-Saharan Africa, using a cluster randomized controlled trial (CRCT), so as to improve proper hand washing, increase knowledge level and also reduce school absenteeism.

DETAILED DESCRIPTION:
A cluster randomized controlled trial (CRCT) design with pre-, mid- and post-interventions and follow-up measures will be randomized into intervention or control groups. A simplified 5-steps hand washing program will be implemented in the intervention group while the control group will continue with their usual practice where schoolchildren do not follow any standard recommended handwashing technique.

ELIGIBILITY:
Inclusion Criteria:

* Schools that have piped tap water source situated in Mzuzu City,
* Private primary schools,
* Children in elementary one and six,
* Written parental consent allowing their child to participate in the study.

Exclusion Criteria:

* Schools without piped tap water source,
* Government primary schools,
* Children whose parents will not give consent.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Proper hand washing | 9 month
  This will be achieved by giving a score to the amount of fluorescents stain on the hand.

SECONDARY OUTCOMES:
Knowledge gain | 9 month
  A quiz will be administered to assess knowledge of school children.

CONTACTS AND LOCATIONS:
Locations (1):
- St John's College of Nursing and Midwifery, Mzuzu, Northern Region, Malawi